CLINICAL TRIAL: NCT04996368
Title: A Randomized Comparison of Two Doses of Tranexamic Acid in Open-Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SGNHC 4
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Drug Use
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The doses of tranexamic acid used during cardiac surgery varies with the institutions that ranges from 10mg/kg to 100mg/kg. This study aims to compare two doses of tranexamic acid, one dose is a conventional dose ( 30mg/kg) and the other is low dose 10mg/kg. Effects of tranexamic acid regarding its effectiveness and side effects profile will be observed. Participants will be randomly selected into two groups ( low dose group and high dose group)
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized into two groups by sealed envelop methods. The primary investigator and participants will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose (10mg/kg) (Active Comparator): The dose of tranexamic acid varies widely ranging from 10mg/kg to 100mg/kg. We are comparing 10mg/kg to conventional 30mg/kg dose. The result of this study will help us to review our current practice.
  Interventions: Drug: Tranexamic acid injection
- high dose or conventional group (30mg/kg) (Active Comparator): dose 30mg/kg regularly use in our center as a prophylaxis for prevention of bleeding before open heart surgery
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — Randomized comparison of two doses of tranexamic acid as prophylactic before start of incision in open heart surgery use for prevention of bleeding.

SUMMARY:
Perioperative bleeding during cardiac surgery is associated with a higher incidence of reoperation and blood transfusion leading to an increase in morbidity and mortality. Coagulopathy is a major cause of excessive bleeding. It is associated with use of cardiopulmonary bypass which activates the intrinsic and extrinsic coagulation pathway, platelet dysfunction and systemic inflammatory response. Increase in duration of cardiopulmonary bypass correlates directly with increase bleeding during cardiac surgery. Antifibrinolytic agents like tranexamic acid has shown promising result in major surgeries and in trauma patients. Current clinical practice guidelines recommended use of tranexamic acid in cardiac surgery. There are wide variations in dose of tranexamic acid ranging from 10mg/Kg to 100mg/kg. The higher dose of this drug is associated with seizures and thromboembolic events including stroke. The objective is to find out the minimal effective dose of tranexamic acid in open-heart surgery.

This is a prospective comparative study among the patients undergoing open heart surgery in Shahid Gangalal National Heart Center, Kathmandu Nepal. The inclusion criteria include patients with age more than 18years, surgery with total cross clamp time more than 60 min. The exclusion criteria are the patients with allergy to tranexamic acid or any of the lysine analogues, history of seizure, chronic homeostasis abnormality, on anticoagulants, severe chronic kidney disease with creatinine clearance less than 30ml/hr, deranged liver function test, total cross clamp time less than 60 min. The sample size was calculated to be 100 including 10% dropout cases. Patients will be randomized into two groups Group H (High dose group) and Group L (Low dose group) with a sealed envelope technique. Low-dose TEA consists of 10 mg/kg bolus administration before incision, followed by1 mg/kg/hr infusion; High-dose TEA consists of a 30 mg/kg bolus followed by a 1mg/kg/hr infusion till the end of surgery. Blood sampling and transfusion will be done as per protocol of Shahid Gangalal National Heart Center. The primary study endpoint was the amount of blood loss during the first 24 hours after surgery. The secondary endpoint was the incidence of overall blood transfusion and hemoglobin concentration on the first postoperative day after surgery. All adverse effects of the drug were noted and were treated as per hospital protocol. Data will be collected using the data collection form (proforma). Collected data will be analyzed by means of spss version 20 for windows. The result will be presented as mean ± SD. The continuous variable will be compared between the two groups by student t test and categorical variables with the chi-square test. A minimum level of significance is maintained at the p-value of <0.05.

DETAILED DESCRIPTION:
Perioperative bleeding is a common complication during cardiac surgery. This is associated with higher incidence of reoperation and blood transfusion increasing morbidity and mortality. [1,2] Coagulopathy is a major cause of excessive bleeding. It is associated with use of cardiopulmonary bypass which activates the intrinsic and extrinsic coagulation pathway, platelet dysfunction and systemic inflammatory response. [3,4] Increase in duration of cardiopulmonary bypass correlates directly with increase bleeding during cardiac surgery. Antifibrinolytic agents like tranexamic acid has shown promising result in major surgeries and in trauma patients. Tranexamic acid blocks reversibly the lysine binding sites of plasminogen. It prevents the activation of plasmin and thus stops lysis of polymerized fibrin.[5] Current clinical practice guidelines recommended use of tranexamic acid in cardiac surgery.[6] The significance for use of this drug is more for the cardiac surgery with higher risk of bleeding like Aortic valve surgery, Coronary artery bypass grafting, redo surgeries and surgery with prolong cardiopulmonary bypass time.[7] However, there is wide variation in dose of tranexamic acid ranging from 10mg/Kg to 100mg/kg.[8] The tranexamic acid use is not free from adverse events. The higher dose of this drug is associated with seizures and thromboembolic events including stroke. [9,10] The objective of this study is to find out the minimal effective dose of tranexamic acid in high-risk open-heart surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18years scheduled for cardiac surgery and requiring CPB
* Surgery with total cross clamp time more than 60 min (Aortic valve surgery, double valve, CABG)

Exclusion Criteria:

* Allergy to tranexamic acid or any of the lysine analogues
* History of seizure
* Chronic homeostasis abnormality, platelet <100000/cumm PT>20sec INR>2
* On anticoagulant
* Severe chronic kidney disease with creatinine clearance less than 30ml/hr
* Deranged liver function test
* Total cross clamp time less than 60 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
amount of blood loss | first 24 hour post operative period
  to compare the amount of blood loss in two group in first 24 hour post operative

SECONDARY OUTCOMES:
blood tranfusion in first 24 hours | first 24 hour post operative period
  To compare total blood products transfused during 24 hours post-operative period
Reoperations for surgical hemostasis | first 24 hour post operative period
  To compare the incidence of reoperations
Adverse drug reactions | first 24 hours
  To Compare the adverse drug reactions between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Gangalal Nationnal Heart Centre, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to anybody. It will be kept confidential. Overall result of the study will be published.

REFERENCES:
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Robich MP, Koch CG, Johnston DR, Schiltz N, Chandran Pillai A, Hussain ST, Soltesz EG. Trends in blood utilization in United States cardiac surgical patients. Transfusion. 2015 Apr;55(4):805-14. doi: 10.1111/trf.12903. Epub 2014 Nov 2. PMID 25363570
- [Background] Biancari F, Mikkola R, Heikkinen J, Lahtinen J, Airaksinen KE, Juvonen T. Estimating the risk of complications related to re-exploration for bleeding after adult cardiac surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2012 Jan;41(1):50-5. doi: 10.1016/j.ejcts.2011.04.023. PMID 21640602
- [Background] Ranucci M, Bozzetti G, Ditta A, Cotza M, Carboni G, Ballotta A. Surgical reexploration after cardiac operations: why a worse outcome? Ann Thorac Surg. 2008 Nov;86(5):1557-62. doi: 10.1016/j.athoracsur.2008.07.114. PMID 19049749